CLINICAL TRIAL: NCT03297554
Title: Healthy Kids Pilot
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed on May 30, 2018 and no participants were enrolled.
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Amanda Staiano, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 2017-044
Record Dates: First submitted 2017-09-18; First posted 2017-09-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- m-health approach (Experimental): See intervention description
  Interventions: Behavioral: m-Health Intervention

INTERVENTIONS:
Behavioral: m-Health Intervention — Parent/child dyads attend remote counseling sessions delivered over Internet-connected device (e.g. smartphone, iPad/tablet, laptop, or desktop computer). A counselor will deliver the lesson, review progress based on the objectively measured data, and provide individualized advice and problem-solving strategies for parent and child. Families will receive weekly contact via smartphone. Each lesson will include an interactive component for parent and child related to healthy eating and active play, as well as an interactive parenting training component. Lessons are based on the family treatment methods that effectively promote child and parent weight loss that is sustained for 10 years (Epstein et al., 1990; Epstein et al., 1981).

SUMMARY:
Up to 30 parent/child dyads will be recruited to participate in an m-Health intervention (delivered over smartphone, iPad/Tablet, or desktop/laptop) to promote healthy behaviors and healthy weight among children and their parents.

ELIGIBILITY:
Inclusion Criteria for Child:

* Have at least one participating parent
* Have a BMI percentile > 85
* Be physically capable of exercise
* Be free of diseases that affect metabolism, body weight, and food intake, including type 1 or type 2 diabetes, HIV/AIDS, and cancer

Inclusion Criteria for Parent:

* Have a smartphone
* Be willing to use the smartphone for the mHealth intervention

Exclusion Criteria for Child:

* Significant cardiovascular disease or disorders via self-report from parent
* Other significant medical problems that would prevent them from engaging in regular physical activity.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Acceptability/feasibility of the mHealth approach | Week 0 to Week 14-16
  Acceptability/feasibility of the mHealth approach will be evaluated by a survey on treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Staiano, PhD, Principal Investigator — Pennington Biomedical Research Center; Corby Martin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Staiano AE, Shanley JR, Kihm H, Hawkins KR, Self-Brown S, Hochsmann C, Osborne MC, LeBlanc MM, Apolzan JW, Martin CK. Digital Tools to Support Family-Based Weight Management for Children: Mixed Methods Pilot and Feasibility Study. JMIR Pediatr Parent. 2021 Jan 7;4(1):e24714. doi: 10.2196/24714. PMID 33410760